CLINICAL TRIAL: NCT02885220
Title: A Randomized Controlled Trial Comparing Goal Directed Versus Conventional Weight Loss Program Post Laparoscopic Sleeve Gastrectomy
Brief Title: Goal Directed Versus Conventional Weight Loss Program
Acronym: Go-Pro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DSRB 2015/00744
Record Dates: First submitted 2016-06-21; First posted 2016-08-31 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Program (Active Comparator): The aim of our study is to determine if a goal directed program improves weight loss outcomes after sleeve gastrectomy. In the conventional weight loss program, patients will only be given their ideal weight to strive toward after surgery. Routine dietary and physiotherapy/exercise counseling are provided and patients would be educated on their ideal weights based on a BMI of 23. The target weight loss over a 12 month period would be 100% excess weight loss.
  Interventions: Other: Conventional Program
- Goal Directed Program (Experimental): For the goal directed program, patients would be given an additional sheet to show expected weight loss goals to strive towards at each consultation after surgery (3, 6, 9 and 12 months post operation). Bariatric patients in this modified program will be counselled prior to laparoscopic sleeve gastrectomy (LSG) and EWL (excess weight loss) targets will be set for patients to achieve at fixed intervals post LSG. These targets are charted in a graph, with the patient's actual weight charted on the graph at each clinic consultation, providing a strong visual aid counselling and motivation.
  Interventions: Other: Goal-directed Program

INTERVENTIONS:
Other: Conventional Program — No scheduled intermediate weight loss goals provided to patient
  Arms: Conventional Program
Other: Goal-directed Program — Scheduled program with intermediate weight loss targets reinforced to patients during follow up.
  Arms: Goal Directed Program

SUMMARY:
The aim of our study is to determine if the goal directed weight loss program improves weight loss versus the conventional weight loss program after laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
The aim of our study is to determine if a goal directed program improves weight loss outcomes after sleeve gastrectomy. Bariatric patients are managed by a multidisciplinary team comprising of bariatric surgeons, dieticians, physiotherapists, and physicians. In the conventional weight loss program, patients were only given their ideal weight to strive toward after surgery. Previous patients undergoing bariatric surgery in the standard program often enquired about the expected excessive weight loss targets after bariatric surgery. This patient driven need led to the development of the goal directed weight loss program. This modified program involves a component of behavioural intervention. Bariatric patients in this modified program will be counselled prior to LSG and EWL targets will be set for patients to achieve at fixed intervals post LSG. These targets are charted on a graph, with the patient's actual weight charted on the same graph at each clinic consultation, providing a strong visual aid to counseling and motivation.

The aim of the study is to recruit 120 patients undergoing laparoscopic sleeve gastrectomy. These patients will be randomized to either the goal directed program or a standard program. Patient demographics, preoperative weight, and post operative weights at 3, 6, 9, 12, 18 and 24 months post laparoscopic sleeve gastrectomy will be collected. Univariate and multivariate analyses will be performed between each group with excess weight loss being the primary endpoint.

Such a trial would allow evaluation to know if the effort spent in implementing a goal directed weight loss program translates to improved weight loss outcomes in bariatric surgery patients. There are no significant risks involved in implementing such a program for our patients. This is based on a retrospective review of patients who have undergone the goal directed program in NUH. If such a program is shown to improve weight loss outcomes post surgery, it could potentially be adopted by bariatric centers worldwide. If the goal directed program is shown to have no bearing on weight loss outcomes, the extra efforts by the bariatric team into implementing such a program could be better directed to other endeavours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having met the indications for laparoscopic sleevel gastrectomy, determined preoperatively by the attending surgeon
2. Age >21 or <65
3. BMI >32.5 and <45
4. Mentally Sound
5. Agreeable to commit to the length of follow up
6. Agreeable for randomization and signed consent form

Exclusion Criteria:

1. No signed consent form
2. Age <21 or >65
3. BMI <32.5 or >45
4. Previous Bariatric surgery
5. Mentally Unsound
6. Unable to commit to follow up schedule
7. Pregnant women or women who are breast-feeding

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2022-09 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Mean excess weight loss | 12 months

SECONDARY OUTCOMES:
Quality of life (SF36 questionaire) | 12 months
Complications and adverse events | 12 months
Remission of co-morbidities | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Locke, E. A. (1996). Motivation through conscious goal setting. Applied and Preventive Psychology, 5(2), 117-124.
- [Background] Wing, R. R. (2002). Behavioral weight control. Handbook of obesity treatment, 2, 301-317.
- [Background] Wadden TA, Foster GD. Behavioral treatment of obesity. Med Clin North Am. 2000 Mar;84(2):441-61, vii. doi: 10.1016/s0025-7125(05)70230-3. PMID 10793651
- [Background] Kim G, Tan CS, Ng JY, Cheng AKS, Rao J, Soe KT, Kong LW, Naseer F, Er PSY, Lomanto D, So JBY, Shabbir A. Goal-directed program after sleeve gastrectomy improves weight loss. Surg Obes Relat Dis. 2016 Mar-Apr;12(3):518-521. doi: 10.1016/j.soard.2015.11.014. Epub 2015 Nov 19. PMID 26944549